CLINICAL TRIAL: NCT05144425
Title: Evaluation of Blood Loss and Pain in TKA With and Without Pneumatic Tourniquet, A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed elbasel abd-elraheem, Assiut medical school ethical review board [assiut], Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Elbasel
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Total Blood Loss
Keywords: total knee arthroplasty
MeSH Terms: conditions — Exsanguination | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): underwent TKA with using pneumatic tourniquet
  Interventions: Procedure: total knee arthroplasty with and without using pneumatic tourniquet
- group B (Placebo Comparator): underwent TKA without using pneumatic tourniquet
  Interventions: Procedure: total knee arthroplasty with and without using pneumatic tourniquet

INTERVENTIONS:
Procedure: total knee arthroplasty with and without using pneumatic tourniquet — The randomization will be performed by a research fellow who will not be involved in patient care. All of the operations will be performed through the medial parapatellar approach by experienced knee surgeons. Drainage system will be used for 48 hours postoperative. In the tourniquet group, the tourniquet will be inflated to a pressure of systolic blood pressure plus 100 mm Hg and will be released after the joint capsule has been closed. hemostasis and then will be wrapped with elastic bandages. In the non-tourniquet group, the tourniquet will be wrapped around the thigh but will not be inflated during the surgery. The criterion for a blood transfusion will set as a hemoglobin (Hb) level of<8 g/dL or patient with symptomatic anemia.

SUMMARY:
The aim of our study is to determine whether the use of a tourniquet during TKA would affect total measured blood loss , operation time, postoperative complications; hemoglobin concentration; limb swelling and postoperative pain.

DETAILED DESCRIPTION:
Tourniquets are widely used in total knee arthroplasty (TKA) . TKA has been reported to be associated with significant blood loss which at times necessitates transfusion. Although the tourniquet is widely used by orthopedic surgeons, its role is controversial . Several studies have shown that using a tourniquet in TKA could reduce the total blood loss, while results from others indicated the opposite . Therefore the relationship between the use of a tourniquet and the total blood loss of patients undergoing TKA is still unclear. The use of a tourniquet is believed to be effective for decreasing intraoperative blood loss and creating a bloodless surgical field, which theoretically would facilitate the cementing technique and other surgical procedures. However, reactive blood flow reaches its peak within five minutes after the tourniquet has been released Complications reported as a consequence of tourniquet application are skin injury [skin abrasions, blisters, breaks , pressure necrosis], nerve injury, post tourniquet syndrome, Deep venous thrombosis, Postoperative pain, wound healing disorders and early infections

ELIGIBILITY:
Inclusion Criteria:

* any patient with knee osteoarthritis undergoing primary total knee arthroplasty

Exclusion Criteria:

1. patients with hemorrhagic disease
2. patient with revision total knee arthroplasty
3. patient with history of vascular thrombosis
4. patients taking anti-platelet agents due to cardiovascular disease
5. patients with hemoglobin level below 10gm/dl

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
amount of perioperative blood loss in ml with and without using tourniquet during TKA | 48hr
  Total measured blood loss will be calculated as the volume of the intraoperative blood loss plus the volume of postoperative visible blood loss from the hemovac drains and will be expressed as mL

SECONDARY OUTCOMES:
post operative pain measured on VAS after TKA with and without using tourniquet | 48hr
  Knee joint pain will be measured on a visual analog scale (VAS) (range, 0-10) pre-operatively and on the 3rd, 5th, 7th and 14th postoperative days [12]. A higher score on the VAS equates to a higher level of pain.
operative time in minutes with and without using tourniquet in TKA | operation time
  operative time in minutes will be calculated and compared the two groups
hemoglobin level in gm/dl preoperative and postoperative | 48hrs
  Hemoglobin level will be measured pre-operatively and after 24hrs and 48 hrs post-operatively. Patients with Hb < 8 g/dl or those who have exhibited symptoms of acute anemia will receive blood transfusion therapy. The amount of blood transfused will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmed Mahran, MD, Study Chair — staff member at assuit university faculty of medicine orthopedic department

REFERENCES:
- [Background] Arthur JR, Spangehl MJ. Tourniquet Use in Total Knee Arthroplasty. J Knee Surg. 2019 Aug;32(8):719-729. doi: 10.1055/s-0039-1681035. Epub 2019 Mar 1. PMID 30822788
- [Background] Nicolaiciuc S, Probst P, von Eisenhart-Rothe R, Burgkart R, Hube R. Modern Total Knee Arthroplasty (TKA): With Or Without a Tourniquet? Surg Technol Int. 2019 Nov 10;35:336-340. PMID 31282982
- [Background] Cai DF, Fan QH, Zhong HH, Peng S, Song H. The effects of tourniquet use on blood loss in primary total knee arthroplasty for patients with osteoarthritis: a meta-analysis. J Orthop Surg Res. 2019 Nov 8;14(1):348. doi: 10.1186/s13018-019-1422-4. PMID 31703706